CLINICAL TRIAL: NCT04165460
Title: Effect of Two Cognitive-Behavioral Interventions on Psychosocial Factors and Quality of Life of Cervical Cancer Patients With Locally-advanced and Advanced Disease
Brief Title: Effect of Two Cognitive-Behavioral Interventions on Cervical Cancer Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Cancerología (Other Government)
Responsible Party: Principal Investigator, Lucely Cetina Pérez, Principal Investigator, National Institute of Cancerología
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 019/026/ICI, CEI/1330/18; INCAN (Other: Instituto Nacional de Cancerología)
Record Dates: First submitted 2019-10-07; First posted 2019-11-18 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Cervical Cancer; Psychological Distress; Coping Skills
Keywords: Cervical cancer; Quality of life; Coping; Distress; Anxiety; Depression; Therapeutic adherence; Sexual Satisfaction
MeSH Terms: conditions — Uterine Cervical Neoplasms; Anxiety Disorders; Depression; Treatment Adherence and Compliance; Orgasm | interventions — Cognitive Restructuring

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- "A" Intervention (Experimental): Psychoeducation, Relaxation, Cognitive Reestructuring and Problem Solving
  Interventions: Other: Psychoeducation; Other: Relaxation; Other: Cognitive Restructuring; Other: Solving Problems
- "B" Intervention (Active Comparator): Psychoeducation, Relaxation
  Interventions: Other: Psychoeducation; Other: Relaxation

INTERVENTIONS:
Other: Psychoeducation — Delivering systematic information about cancer, oncological treatment and efficient coping strategies.
Other: Relaxation — Teaching the patient in diaphragmatic breathing retraining and passive relaxation with guided imagination.
Other: Cognitive Restructuring — Teaching the patient to identify dysfunctional cognitions about cancer and oncological treatment that trigger maladaptive emotions and behavior. Then, focus in generating alternative thoughts through contrast with empirical reality based on the Beck Model.
  Arms: "A" Intervention
Other: Solving Problems — To generate alternative solutions to practical problems based on the model described by Nezu.
  Arms: "A" Intervention

SUMMARY:
Cancer represents the second cause of death in general population worldwide and according to statistics, it is expected to increase in the next 20 years. Cervical cancer is the fourth cause of morbidity and mortality among women around the world. Late diagnosis and treatment indices several emotional reactions in patients leading to psychological disorders with an impact in quality of life. Anxiety and depression are the most frequent emotional reactions in cancer patients, which may vary depending on psychosocial factors such as coping and family support, mostly provided by the primary caregiver. Despite the high psychological morbidity in cancer patients, it is estimated that, among those patients needing psychological support, only 10% receive such interventions. A growing interest on psychological interventions in oncology has increased in the last 40 years, however, scarce investigations have been performed, especially in cervical cancer patients. The Cognitive-Behavioral Therapy has proven to be beneficial in general cancer population decreasing the psychological symptoms and improving the quality of life. Thus, the aim of this study is to evaluate the effect of two Cognitive-Behavioral psychological interventions on anxiety, depression, coping, therapeutic adherence, sexual satisfaction and quality of life of cervical cancer patients with locally-advanced and advanced disease attended at the National Cancer Institute from Mexico. Psychological intervention will be provided during ten weekly sessions including psychoeducation, relaxation, cognitive restructuring and problem solving with a pretest, posttest performed one week after intervention, and finally a follow up after three months after finishing the psychological intervention.

DETAILED DESCRIPTION:
Cervical cancer is the fourth cause of morbidity and mortality worldwide, being one of the most important threats to women's health. More than 83,000 women were diagnosed with cervical cancer and 36,000 died in the Region of the Americas in 2012. This phenomenon will increase by 45% for 2030.

During the natural history of Cervical cancer, and as a consequence of therapeutic approaches, a certain proportion of the patients may have emotional reactions leading to psychological disorders, as severe as those disease complications, which also deteriorate their quality of life. The most frequent reactions are anxiety and depression. These may vary depending on different psychosocial factors, including coping and social support, mostly provided by the Primary Caregiver, who has a fundamental role in hospital and home care, helping on therapeutic adherence.

Therapeutic adherence is essential in order to obtain optimal results of the given oncological treatment, representing a mediating variable with important implications for survival, disease progression and in the improving of quality of life.

Response to treatment has been widely evaluated by tumor size, OS and DFS. Nevertheless, in the past tree decades the evaluation of Quality of Life has risen as an indicator of therapeutic response. Quality of life is an indicator that measures the general well-being of the patients according to the overall effects of the oncological treatments. Scientific evidence reports that cervical cancer survivors may have a worst quality of life as well as other physical and emotional symptoms than those observed in other cancer populations. Hence, it is necessary to focus on psychological interventions aimed to improve the quality of life and to decrease the psychological morbidity in cervical cancer patients.

During the last four decades a special interest in psychosocial interventions in oncology population has risen, establishing that Cognitive-Behavioral Therapy is beneficial in the reduction of physical and emotional symptoms of patients, promoting the adaptive coping and improving the quality of life.

Few evidences exist about psycho-social factors prevalence on gynecological cancer patients. The current available studies have grouped different types of gynecological cancer including breast, ovary, endometrium and vulva, but cervical cancer has been included only in a small proportion of those studies producing a certain degree of bias at the time of interpreting the results. Moreover, most of the studies has focused in breast and ovarian cancer patients. However, it has been proposed the existence of differences in psychological morbidity in women with cervical cancer, therefore is essential to focus our efforts in this particular population due to its high morbidity and mortality.

Hypothesis Patients with locally advanced and advanced cervical cancer receiving "A" psychological intervention will have a greater decrease in anxiety, depression, better coping responses, sexual satisfaction, therapeutic adherence and quality of life compared with the "B" psychological intervention.

The general aim of this study is to evaluate the effect of two cognitive-behavioral interventions on psycho-social factors and quality of life of cervical cancer patients with locally advanced and advanced disease.

Specific objectives:

1. To identify and to compare the degree of the psychosocial variables: anxiety, depression, coping responses, therapeutic adherence and sexual satisfaction at different evaluation phases (pre-intervention, post-intervention and follow-up) in cervical cancer patients.
2. To evaluate and to compare the health-related quality of life perceived at different evaluation phases (pre-intervention, post-intervention and follow-up) in cervical cancer patients.

Exploratory objectives:

1. To evaluate the degree of anxiety, depression, quality of life and the presence of Caregiver Burden Syndrome in primary caregivers before the psychological treatment given to cervical cancer patients.
2. To evaluate the association between psychological variables of the primary caregiver and the emotional distress and quality of life of their locally advanced and advanced cervical cancer patients.

METHODS

Study Design: This a prospective, experimental, longitudinal, open and randomized study

Study population: patients will be divided into two treatment groups ("A" and "B") for pre-intervention, post-intervention and a three months follow-up evaluation treated at the National Cancer Institute from Mexico.

Sample size:

According to the criteria of two proportions, a sample of 92 cervical cancer patients (two intervention groups) and their matched primary caregivers (92) was obtained.

Statistical analysis:

The processing and analysis of the database will be carried out with the SPSS version 22.0® package for Microsoft.

* Univariate analysis will be carried out to describe the study population. Descriptive statistics will be used to obtain measures of central tendency and dispersion, for continuous variables depending on their distribution, mean and standard deviation (parametric) or median and interquartile range (non-parametric) may be reported. For qualitative variables, the distribution of absolute and relative frequencies will be reported.
* Group homogeneity analysis: the general characteristics of the patients in both intervention groups will be evaluated to asses the balance and homogeneity. For quantitative variables t-Student of independent samples or U of Mann-Whitney will be used. For qualitative variables Chi-Square or Chi-Square trends will be used.
* To estimate the change in the variables of interest throughout the measurements in both intervention groups, ANOVA analysis of repeated measures or Friedmand will be carried out.
* To determine the clinical intra-subject changes, an analysis of individual replicates will be performed analyzing the pre-intervention, post-intervention and after three-month follow-up evaluation.

Procedure:

Patients affiliated to the MICAELA Program referred to the Psychooncology service will be considered as candidates for the study.

Informed consent obtention: after reading the Informed Consent, patients will be informed that their participation will consist on answering questionnaires for psychological assessment and psychological attention, if required. If the patient agree to participate, she will sign the Informed Consent document. A semi-structured interview will be applied to obtain socio-demographic and familiar psycho-pathological disorders history. Then, psychometric instruments will be applied.

Patients who are detected with distress or maladaptive coping will be randomized to one of the two interventions groups.

There will be scheduled ten weekly sessions of one hour approximately in with "A" Intervention or "B" Intervention will be applied according the group assigned by randomization. Then, patients will be scheduled for psychological treatment appointments and for evaluation after finishing treatment.

Ethical considerations:

Participants will be informed about details regarding the study, through the Informed Consent process. Patients that desire to participate will express their willingness with the sign of the Informed Consent document. Patients could leave the study at any time when desire.

The study will be conducted according to the ethical principles established in the documents adopted by the international community as declared at the Good Clinical Practices, the Nuremberg Code, the Declaration of Helsinki as well as the Guide of Good Clinical Practices of the Conference Harmonization International and anyone who represents the greatest protection for the individual.

According to the regulations of the General Health Law on Health Research, the second title on the Ethical Aspects of Research in Human Beings, Chapter I, Article 17, paragraph III, the proposed interventions on this study are considered as risk-free.

Protocol and Informed Consent have been approved by Institutional Research and the Ethics Committees.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS:

  * Affiliated to the MICAELA (Modelo Integral para el Cáncer Cervicouterino Localmente Avanzado y Avanzado) program
  * Ability to understand the study and to provide signed informed consent
  * Diagnosed with locally advanced and advanced cervical cancer
  * Patients newly diagnosed or with recurrence about to start treatment
  * Patients with moderate or severe anxiety, and/or depression symptoms or maladaptive coping
* PRIMARY CAREGIVERS:

  * Relatives, acquaintance or friends reported to be the principal caregiver of the patient
  * Relatives, acquaintance or friends who do not perceived economic remuneration for taking care of the patient

Exclusion Criteria:

* PATIENTS:

  * Patients with psychological or psychiatric treatment or who received previous mental-health treatment.
  * Patients with any alteration of the Central Nervous System
  * Patients with moderated or severe cognitive impairment
  * Patients under palliative care or in terminal phase
* PRIMARY CAREGIVERS

  * Caregivers with severe hearing and/or visual problems
  * Caregivers with a professional or technical training in patient care

Elimination criteria Patients referred to palliative care

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2020-03-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Anxiety and Depression | Six months
  Change in Hospital Anxiety and Depression Scale total score and in the two Subescales
  The Hospital Anxiety and Depression Scale (HADS-M) for Mexican patients. HADS was especially designed to detect anxiety and depression states of patients with chronic diseases. HADS-M is a HADS-modified version that has been validated in an oncological sample of patients in Mexican population. HADS-M comprises 12 items measured in a 0-3-point Likert scale, divided into two subescales, one for depression and one for anxiety. The validated version in Mexico has an internal consistency of alpha= 0.86 for global scale, and 0.79 for depression and 0.80 for anxiety subscales. Compared to other instruments, it has sensitivity to detect therapeutic changes associated to psychological interventions. The subscales score is categorized in without (0-5), low (6-8), moderate (9-11), and severe (12 or more) anxiety or depression.
Change in coping style | Six months
  Change in the Brief COPE-17 Inventory subescales scores
  The Brief COPE Inventory (COPE-17). Is a brief version of the COPE Inventory (Carver, et al., 1989). It has 17 items measured in a 0-3 point Likert scale, to evaluate coping strategies, that are grouped in seven subescales (planning, self-distraction, humor, seeking for social support, substance use, emotional-religious-spiritual support and self-blame). COPE-17 determines two primary coping styles either as approach coping or avoidant coping. It was adapted and validated in Mexico on a breast cancer population (Ornelas, et al., 2013), obtaining an internal alpha consistency of 0.70 either for the general scale and for each subescale. Avoidant Coping is characterized by the subscales of self-distraction, substance use and self-blame. Approach Coping is characterized by the subscales of planning and seeking for social support. Humor and Emotional-Religious-spiritual are neither Approach nor Avoidance coping.
Change in general quality of life for cancer patients: EORTC QLQ-C30 v3, in spanish | Six months
  Change in quality of life summary score of The European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30).
  The EORTC QLQ-C30 questionnaire evaluates the quality of life in oncological population, is composed of both multi-item and single-item measures. It has 30 items, including nine scales: five functional scales (physical, role, emotional, cognitive and social functioning), three symptom scales (fatigue, pain and nausea / vomiting) and one global health status/QoL scale. Six single items are also included (Dyspnea, Insomnia, Appetite loss, Constipation, Diarrhea and Financial difficulties). A high score for all functional and global health/QoL scales represents a high/healthy level of functioning/high QoL, whereas a high score for a symptom scale/item represents a high level of symptoms/problems. The QLQ-C30 was validated in mexican population, obtaining a Crombach's coefficient of 0.7 (Oñate-Ocaña, et al, 2009).
Change in quality of life for cervical cancer patients: EORTC QLQ-CX 24 | Six months
  Change in quality of life summary score and subescales using The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Cervical Cancer Module (EORTC QLQ-CX24).
  The EORTC QLQ-CX24 is the supplementary module of the QLQ-C30 aimed to evaluate quality of life of cervical cancer patients. It consists of 24 items divided in three multi-item scales to assess symptoms experience (gastrointestinal and genitourinary), body image and sexual/vaginal functioning, and six single items to assess lymphedema, peripheral neuropathy, menopausal symptoms, sexual worry, sexual activity and sexual enjoyment. The last five questions are answered only by patients with an active sex life. Higher scores are equivalent to worse or more symptoms, except for items 49 and 54 (higher score indicates better quality of life). The responses are in a 4-point Likert scale. There is a Spanish version used in Mexican population that was provided by EORTC to use in this study.
Changes in sexual satisfaction in women treated for cervical cancer | Six months
  Changes in Screening Questionnaire aimed to identify sexual satisfaction in women treated for cervical cancer Screening questionnaire aimed at identifying sexual satisfaction in women treated for cervical cancer. To explore sexual activity and cognitive distortions about sexuality during and after oncological treatment, with 20 questions in a dichotomous yes/no response. It was developed for this study as part of the semi-structured screening interview in order to determine the cognitions that generate emotional distress and affectation in the quality of life.
Changes in the Factors related to therapeutic adherence | Six months
  Changes in the Factors related to therapeutic adherence in cancer patients Scale subscales scores Scale to assess factors related to therapeutic adherence in cancer patients (Urzúa et al., 2012). This scale consists in 20 items measured in a 1-4 point likert scale, it evaluates three factors that may affect the therapeutic adherence of patients to oncological treatment. It has three subescales: a) Expectations and personal tools to face the disease, b) Beliefs about the treatment and c) Perceived effects of the treatment. It was developed especially for oncological population with an internal consistency of alpha=0.96 in the global scale and 0.9, 0.93 and 0.91 for the three subscales.

SECONDARY OUTCOMES:
Physiological changes in blood pressure | Two months
  Quantitative Changes in the records of physiological measures in which blood pressure (mmHg) are recorded before and after performing the training relaxation exercises.
Physiological changes in temperature | Two months
  Quantitative Changes in the records of physiological measures in which temperature (Celsius degrees) are recorded before and after performing the training relaxation exercises.
Physiological changes in heart rate | Two months
  Quantitative Changes in the records of physiological measures in which heart rate (beats/min) are recorded before and after performing the training relaxation exercises.
Physiological changes in breathing rate | Two months
  Quantitative Changes in the records of physiological measures in which breathing rate (breaths/minute) are recorded before and after performing the training relaxation exercises.
Maladaptive thoughts changes | During each Cognitive Reestructuring training session
  Qualitative Changes of automatic thoughts during Cognitive Restructuring Technique will be recorded in order to promote "alternative thoughts" according to the Beck Theory for Cognitive Restructuring.
Correlation of anxiety, depression, caregiver burden syndrome and quality of life | at pretest
  Correlation of the total scores of anxiety, depression, caregiver burden syndrome and quality of life evaluated in the primary Caregiver with the variables of anxiety, depression, coping adherence and quality of life of cervical cancer patients

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Salazar, MSc, Study Chair — National Cancer Institute from Mexico
Locations (1):
- Instituto Nacional de Cancerologia, Mexico City, Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] Die Trill M. Anxiety and sleep disorders in cancer patients. EJC Suppl. 2013 Sep;11(2):216-24. doi: 10.1016/j.ejcsup.2013.07.009. No abstract available. PMID 26217130
- [Background] Mitchell AJ, Chan M, Bhatti H, Halton M, Grassi L, Johansen C, Meader N. Prevalence of depression, anxiety, and adjustment disorder in oncological, haematological, and palliative-care settings: a meta-analysis of 94 interview-based studies. Lancet Oncol. 2011 Feb;12(2):160-74. doi: 10.1016/S1470-2045(11)70002-X. Epub 2011 Jan 19. PMID 21251875
- [Background] Henriksson MM, Isometsa ET, Hietanen PS, Aro HM, Lonnqvist JK. Mental disorders in cancer suicides. J Affect Disord. 1995 Dec 24;36(1-2):11-20. doi: 10.1016/0165-0327(95)00047-x. PMID 8988260
- [Background] Spiegel D, Giese-Davis J. Depression and cancer: mechanisms and disease progression. Biol Psychiatry. 2003 Aug 1;54(3):269-82. doi: 10.1016/s0006-3223(03)00566-3. PMID 12893103
- [Background] Massie MJ. Prevalence of depression in patients with cancer. J Natl Cancer Inst Monogr. 2004;(32):57-71. doi: 10.1093/jncimonographs/lgh014. PMID 15263042
- [Background] Jadoon NA, Munir W, Shahzad MA, Choudhry ZS. Assessment of depression and anxiety in adult cancer outpatients: a cross-sectional study. BMC Cancer. 2010 Oct 29;10:594. doi: 10.1186/1471-2407-10-594. PMID 21034465
- [Background] Hinz A, Krauss O, Hauss JP, Hockel M, Kortmann RD, Stolzenburg JU, Schwarz R. Anxiety and depression in cancer patients compared with the general population. Eur J Cancer Care (Engl). 2010 Jul;19(4):522-9. doi: 10.1111/j.1365-2354.2009.01088.x. Epub 2009 Dec 17. PMID 20030697
- [Background] Dauchy S, Dolbeault S, Reich M. Depression in cancer patients. EJC Suppl. 2013 Sep;11(2):205-15. doi: 10.1016/j.ejcsup.2013.07.006. No abstract available. PMID 26217129
- [Background] Pfaendler KS, Wenzel L, Mechanic MB, Penner KR. Cervical cancer survivorship: long-term quality of life and social support. Clin Ther. 2015 Jan 1;37(1):39-48. doi: 10.1016/j.clinthera.2014.11.013. PMID 25592090
- [Background] Manne SL, Virtue SM, Ozga M, Kashy D, Heckman C, Kissane D, Rosenblum N, Morgan M, Rodriquez L. A comparison of two psychological interventions for newly-diagnosed gynecological cancer patients. Gynecol Oncol. 2017 Feb;144(2):354-362. doi: 10.1016/j.ygyno.2016.11.025. Epub 2016 Nov 23. PMID 27887806
- [Background] Moorey S, Frampton M, Greer S. The Cancer Coping Questionnaire: a self-rating scale for measuring the impact of adjuvant psychological therapy on coping behaviour. Psychooncology. 2003 Jun;12(4):331-44. doi: 10.1002/pon.646. PMID 12748971
- [Background] Watson M, Greer S, Young J, Inayat Q, Burgess C, Robertson B. Development of a questionnaire measure of adjustment to cancer: the MAC scale. Psychol Med. 1988 Feb;18(1):203-9. doi: 10.1017/s0033291700002026. PMID 3363039
- [Background] van Laarhoven HW, Schilderman J, Bleijenberg G, Donders R, Vissers KC, Verhagen CA, Prins JB. Coping, quality of life, depression, and hopelessness in cancer patients in a curative and palliative, end-of-life care setting. Cancer Nurs. 2011 Jul-Aug;34(4):302-14. doi: 10.1097/NCC.0b013e3181f9a040. PMID 21116179
- [Background] Valencia MC, Meza-Osnaya G, Perez-Cruz I, Cortes-Campero N, Hernandez-Ovalle J, Hernandez-Paredes P, Juarez-Romero K, Chino-Hernandez B, Romero-Figueroa MS. [Factors involved in the burden of the primary caregiver of cancer patients]. Rev Calid Asist. 2017 Jul-Aug;32(4):221-225. doi: 10.1016/j.cali.2016.11.003. Epub 2017 Mar 8. Spanish. PMID 28284516
- [Background] Puts MTE, Tu HA, Tourangeau A, Howell D, Fitch M, Springall E, Alibhai SMH. Factors influencing adherence to cancer treatment in older adults with cancer: a systematic review. Ann Oncol. 2014 Mar;25(3):564-577. doi: 10.1093/annonc/mdt433. Epub 2013 Nov 26. PMID 24285020
- [Background] Osann K, Hsieh S, Nelson EL, Monk BJ, Chase D, Cella D, Wenzel L. Factors associated with poor quality of life among cervical cancer survivors: implications for clinical care and clinical trials. Gynecol Oncol. 2014 Nov;135(2):266-72. doi: 10.1016/j.ygyno.2014.08.036. Epub 2014 Sep 3. PMID 25192629
- [Background] Redd WH, Silberfarb PM, Andersen BL, Andrykowski MA, Bovbjerg DH, Burish TG, Carpenter PJ, Cleeland C, Dolgin M, Levy SM, et al. Physiologic and psychobehavioral research in oncology. Cancer. 1991 Feb 1;67(3 Suppl):813-22. doi: 10.1002/1097-0142(19910201)67:3+3.0.co;2-w. PMID 1986851
- [Background] Barton-Burke M, Gustason CJ. Sexuality in women with cancer. Nurs Clin North Am. 2007 Dec;42(4):531-54; vi. doi: 10.1016/j.cnur.2007.08.001. PMID 17996754
- [Background] Baider L, Peretz T, Hadani PE, Koch U. Psychological intervention in cancer patients: a randomized study. Gen Hosp Psychiatry. 2001 Sep-Oct;23(5):272-7. doi: 10.1016/s0163-8343(01)00158-x. PMID 11600169
- [Background] Hopko DR, Bell JL, Armento M, Robertson S, Mullane C, Wolf N, Lejuez CW. Cognitive-behavior therapy for depressed cancer patients in a medical care setting. Behav Ther. 2008 Jun;39(2):126-36. doi: 10.1016/j.beth.2007.05.007. Epub 2007 Oct 31. PMID 18502246
- [Background] Goerling U, Foerg A, Sander S, Schramm N, Schlag PM. The impact of short-term psycho-oncological interventions on the psychological outcome of cancer patients of a surgical-oncology department - a randomised controlled study. Eur J Cancer. 2011 Sep;47(13):2009-14. doi: 10.1016/j.ejca.2011.04.031. Epub 2011 May 24. PMID 21612912
- [Background] de la Torre-Luque A, Gambara H, Lopez E, Cruzado JA. Psychological treatments to improve quality of life in cancer contexts: A meta-analysis. Int J Clin Health Psychol. 2016 May-Aug;16(2):211-219. doi: 10.1016/j.ijchp.2015.07.005. Epub 2015 Aug 29. PMID 30487864
- [Background] Rehse B, Pukrop R. Effects of psychosocial interventions on quality of life in adult cancer patients: meta analysis of 37 published controlled outcome studies. Patient Educ Couns. 2003 Jun;50(2):179-86. doi: 10.1016/s0738-3991(02)00149-0. PMID 12781933
- [Background] Manne SL, Rubin S, Edelson M, Rosenblum N, Bergman C, Hernandez E, Carlson J, Rocereto T, Winkel G. Coping and communication-enhancing intervention versus supportive counseling for women diagnosed with gynecological cancers. J Consult Clin Psychol. 2007 Aug;75(4):615-628. doi: 10.1037/0022-006X.75.4.615. PMID 17663615
- [Background] Galindo-Vazquez O, Benjet C, Cruz-Nieto MH, Rojas-Castillo E, Riveros-Rosas A, Meneses-Garcia A, Aguilar-Ponce JL, Alvarez-Avitia MA, Alvarado-Aguilar S. Psychometric properties of the Zarit Burden Interview in Mexican caregivers of cancer patients. Psychooncology. 2015 May;24(5):612-5. doi: 10.1002/pon.3686. Epub 2014 Sep 29. No abstract available. PMID 25263699
- [Background] Moher D, Schulz KF, Altman DG. The CONSORT statement: revised recommendations for improving the quality of reports of parallel-group randomised trials. Lancet. 2001 Apr 14;357(9263):1191-4. PMID 11323066
- See also: Organización Mundial de la Salud. Cáncer. Nota descriptiva — https://www.who.int/es/news-room/fact-sheets/detail/cancer
- See also: Instituto Nacional de Estadística y Geografía. "Estadísticas a propósito del… Día mundial contra el cáncer (4 de febrero)". Datos nacionales. — http://www.diputados.gob.mx/sedia/biblio/usieg/comunicados/salud2.pdf
- See also: Stewart B, Wild C. World Cancer Report, [monografía en internet]. Ginebra: WHO-OMS-IARC; 2014 — http://iarc.fr/wp-content/uploads/2019/03/brochureWCR2019-web.pdf
- See also: Olivares M. Aspectos psicológicos en el cáncer ginecológico. Avances en Psicología Latinoamericana. 2004;22:29-48. — https://www.redalyc.org/pdf/799/79902205.pdf
- See also: Almanza-Muñoz J, Holland J. Psico-oncología: estado actual y perspectivas futuras. Revista del Instituto Nacional de Cancerología. 2000; 43(3) 196-206. — https://www.medigraphic.com/pdfs/cancer/ca-2000/ca003k.pdf
- See also: Hernández M, Cruzado J. La atención psicológica a pacientes con cáncer: de la evaluación al tratamiento. Clínica y Salud. 2013; 24:1-9. — https://scielo.isciii.es/pdf/clinsa/v24n1/original1.pdf
- See also: Pousa R, Miguelez A, Hernández B, González T, Gaviria M. Depresión y cáncer: una revisión orientada a la práctica clínica. Revista Colombiana de Cancerología. 2015; 47:1-7 — http://www.scielo.org.co/pdf/rcc/v19n3/v19n3a06.pdf
- See also: Rojas O, Fuentes C, Robert V. Psicooncología en el Hospital General. Alcances en depresión y cáncer. Rev. Med. Clin. Condes. 2017;28:450-459. — https://doi.org/10.1016/j.rmclc.2017.05.017
- See also: Barrohilhet S, Forjaz MJ, Garrido LE. Conceptos, teorías y factores psicosociales en la adaptación al cáncer. Actas Especiales de Psiquiatría. 2005; 33:390-397. — http://www.cuidadospaliativos.org/uploads/2010/05/Conceptos,%20teor%C3%ADas%20y%20factores%20psicosociales%20en%20la%20adaptaci%C3%B3n%20al%20c%C3%A1ncer.pdf
- See also: Rangel-Domínguez NE, Ascencio-Huertas L, Ornelas-Mejorada RE, Allende-Pérez SR, Landa-Ramírez E y Sánchez-Sosa JJ. Efectos de la solución de problemas sobre los comportamientos de autocuidado de cuidadores de pacientes oncológicos en fase paliativa: u — https://cuidadospaliativos.org/uploads/2020/12/Asencio%20Solucion%20de%20Problemas.pdf
- See also: Galindo VO, Rojas CE, Ascencio HL, Meneses GA, Aguilar PJL, Opsico-lvera ME et al. Guía de práctica clínica para la atención oncológica del cuidador primario informal de pacientes con cáncer. Psicooncología. 2015; 12(1): 87-104. — https://revistas.ucm.es/index.php/PSIC/article/view/48906/45632
- See also: Organización Mundial de la Salud (OMS). Defining Adherence. En: OMS. (2003). Adherence to long-term therapies. Evidence for action. Switzerland: World Health Organization. 2003; 3-9. — http://apps.who.int/iris/bitstream/handle/10665/42682/9241545992.pdf;jsessionid=FCF9F14E637769CD259A34D351F5AD31?sequence=1
- See also: Palacios-Espinosa X, Vargas-Sterling LP. Adherencia a la quimioterapia y radioterapia en pacientes oncológicos: Una revisión de la literatura. Psicooncología, 2011:2-3. — http://apps.who.int/iris/bitstream/handle/10665/42682/9241545992.pdf;jsessionid=FCF9F14E637769CD259A34D351F5AD31?sequence=1
- See also: Urzúa MA, Marmolejo CA, Barr DC. Validación de una escala para evaluar factores vinculados a la adherencia terapéutica en pacientes oncológicos. Universitas Psychologica. 2012;11(2):587-598. — http://www.scielo.org.co/pdf/rups/v11n2/v11n2a20.pdf
- See also: Sánchez R, Ballesteros M, Gómez AA. Medición de la calidad de vida en ensayos clínicos de pacientes con cáncer. Un estudio bibliométrico. Revista Colombiana de Cancerología. 2009; 13(1):29-34. doi: 10.1016/S0123-9015(09)70149-0. — https://www.redalyc.org/pdf/804/80401403.pdf
- See also: Arraras JI, Martínez M, Manterota A, Laínez N. La evaluación de la calidad de vida del paciente oncológico. El grupo de calidad de vida de la EORTC. Psicooncología. 2004; 1(1):87-98. — https://scielo.isciii.es/scielo.php?script=sci_arttext&pid=S1137-66272011000100002
- See also: Pinzón FCE. Cuestionamientos y requerimientos en la investigación de la calidad de vida en oncología. Revista Colombiana de Psiquiatría. 2010; 39(1):153-167. — https://www.elsevier.es/es-revista-revista-colombiana-psiquiatria-379-avance-resumen-cuestionamientos-requerimientos-investigacion-calidad-vida-S0034745014602420
- See also: Galindo VO, Bejet C, Juárez GF, Rojas CE, Riveros RA, Aguilar PJL et al. Propiedades psicométricas de la Escala Hospitalaria de Ansiedad y Depresión (HADS) en una población de pacientes oncológicos mexicanos. Salud Mental. 2015;38 (4):253-258. — https://doi.org/10.25009/pys.v32i2.2752
- See also: Galindo VO, Meneses GA, Herrera GA, Caballero TR, Aguilar PJL.Escala Hospitalaria de Ansiedad y Depresión (HADS) en cuidadores primarios informales de pacientes con cáncer: propiedades psicométricas. Psicooncología. 2015; 12(2-3) 383-392. — https://www.scielo.org.mx/scielo.php?script=sci_arttext&pid=S0185-33252015000400253